CLINICAL TRIAL: NCT03102619
Title: Wireless Assessment of Respiratory and Circulatory Distress; A Pilot Study
Acronym: WARD
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Camilla Lundgreen Duus, Research Assistant, Bispebjerg Hospital
Other Study IDs: Bispebjerg Hospital
Record Dates: First submitted 2017-03-24; First posted 2017-04-06 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Abdominal Cancer; Postoperative Complications; Respiratory Complication; Circulatory; Complications
Keywords: Wireless monitoring; Postoperative complications; Vital parameters; Continuous monitoring
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Postoperative observation of patients is based on the Early Warning Score (EWS). By using continuous wireless monitoring of vital parameters it may be possible to predict the risk of complications after abdominal cancer surgery. The object of this pilot study is to test the equipment and methods for the next phases. Patients will be monitored for 4 days postoperatively and data is analyzed retrospectively. Vital parameters are monitored with ECG, blood pressure monitor and pulseoximetry.

In the analysis the investigators will compare the results from the continuous monitoring to the measurements made by the nurses and registered in the EWS. The primary outcomes for the pilot study are the frequency of measurements resulting in a single parameter score of 3 according to the EWS algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer of either esophagus, stomach, pancreas, liver, colon or rectum.
* Elective surgery with curative intention at Bispebjerg Hospital or Rigshospitalet in Copenhagen, Denmark.
* Estimated duration of surgery > 2 hours
* > 65 years
* Preoperative ECG showing sinus rhythm
* No treatment limitations
* Fit to receive optimized care according to the regimens on the given wards

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing major abdominal cancer surgery with a curative intention at either Bispebjerg Hospital or Rigshospitalet.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Heart rate resulting in a single parameter score of 3 according to EWS algorithm | The patients are monitored for 4 days
  All data from the monitoring will be analyzed using the thresholds from the EWS algorithm and will be sorted into relevant categories. The following thresholds are used:
  Bradycardia: pulse < 41 bpm Tachycardia: pulse > 130 bpm
Respiration rate resulting in a single parameter score of 3 according to EWS algorithm | The patients are monitored for 4 days
  Bradypnea: < 9 breaths/min Tachypnea: > 24 breaths/min
Blood pressure resulting in a single parameter score of 3 according to EWS algorithm | The patients are monitored for 4 days
  Hypotension: Systolic blood pressure < 91 mmHg Hypertension: Systolic blood pressure > 219 mmHg
Blood oxygen saturation resulting in a single parameter score of 3 according to EWS algorithm | The patients are monitored for 4 days
  Hypoxemia: arterial oxygen saturation < 92 %

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Meyhoff, MD, PhD, Study Chair — Bispebjerg Hospital; Eske K Aasvang, MD, DMSci, Study Chair — Rigshospitalet, Denmark; Helge B Dissing, PhD, Study Chair — Technical University of Denmark; Camilla L Duus, MB, Principal Investigator — Bispebjerg Hospital
Locations (2):
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Bispebjerg Hospital, Copenhagen